CLINICAL TRIAL: NCT02559765
Title: Current Access to, Use and Perceived Efficacy of Physiotherapy and Rehabilitation Services by People With Progressive Multiple Sclerosis: a Survey of People With Progressive Multiple Sclerosis Via the UK MS Register.
Brief Title: Access, Use and Opinions of Physiotherapy and Rehabilitation Services of People With Progressive MS in the UK.
Status: Completed | Type: Observational
Sponsor: University of Glasgow (Other)
Collaborators: NHS Ayrshire and Arran (Other); AKM (Other)
Responsible Party: Principal Investigator, Evan Campbell, Research physiotherapist, University of Glasgow
Other Study IDs: 200140102
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Progressive Multiple Sclerosis
Keywords: physiotherapy; progressive multiple sclerosis; rehabilitation; rehabilitation services
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This survey will investigate the views of people with progressive MS in terms of physiotherapy services. In particular the study will examine the proportion of people with progressive MS on the MS register who use physiotherapy services, how worthwhile they think it is for them and how they would like their physiotherapy to be delivered. This survey will also explore how physiotherapy services for people with progressive MS varies across the UK and what other types of rehabilitation services are currently used by people with progressive MS.

DETAILED DESCRIPTION:
Multiple Sclerosis has three main forms: Relapsing Remitting MS (RRMS), Primary Progressive MS (PPMS) and Secondary Progressive MS (SPMS) as well as a rarer form called Progressive Relapsing MS (PRMS).

In cases of RRMS an individual will have periods of worsened symptoms followed by periods of remission. During remission the individual may make a full recovery or be left with some residual impairment. In both PPMS and SPMS an individual will have continuous worsening symptoms with a gradual increase in disability with little or no transient recovery. An individual with PRMS will have the continuous worsening of disability seen in both PPMS and SPMS coupled with occasional relapses as seen in RRMS.

Currently 15% of those with MS are diagnosed as PPMS, 5% are diagnosed with the rarer form of PRMS and approximately 80% are diagnosed with RRMS. However, approximately 65% of those with RRMS will go on to develop SPMS. This means that approximately 72% of all individuals with MS will be in a progressive phase of the disease at some point in their life.

Whilst there are disease modifying drugs available for those with RRMS there are currently limited pharmacological treatments available for those with the progressive forms of the disease. Physiotherapy and rehabilitation services are often used by people with progressive MS and access to these are part of the current NICE guidelines for the management of MS. Whilst physiotherapy and rehabilitation services are used by people with progressive MS there is currently no research investigating how many people with progressive MS use these services, who provides them, how they are delivered, how effective the recipient feels the treatment is and how they would like their service to be delivered. In addition the Progressive MS Alliance has highlighted progressive MS and symptom management and rehabilitation as an under-researched area.

The UK MS Register is funded by the MS Society and operated by the health informatics department within the College of Medicine at Swansea University. People with MS can sign up to the register and answer pre-set questionnaires online. The purpose of the Register is to be a longitudinal research database collecting routine data every three months as well as conducting individually commissioned cross sectional studies. It currently has over 11,000 members and over 2,200 of those registrants have a progressive form of MS. Not only is this is the first study with the UK MS register to focus on people with progressive forms of MS but also the first to focus on physiotherapy services.

This is a unique opportunity to access this patient group across a large geographical region and gain an insight into how physiotherapy and rehabilitation services are used, delivered and perceived. The outcome of this research has the potential to inform future physiotherapy interventions and rehabilitation guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Have a form of progressive MS
* Be registered on the UK MS Register

Exclusion Criteria:

* Have relapsing remitting MS
* Be under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with progressive multiple sclerosis and registered on the UK MS Register
Sampling Method: Non-Probability Sample
Enrollment: 1298 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with access to physiotherapy for their MS. Questionnaire | three months
  Questionnaire has the following options: yes, no. Participant may choose one.
Number of participants that use physiotherapy for their MS. Questionnaire | three months
  Questionnaire has the following options: yes, no. Participant may choose one.
What is the participants' perceived efficacy of physiotherapy for their MS? Questionnaire | three months
  Nominal scale of: very harmful, harmful, neither harmful nor beneficial, beneficial, very beneficial Participant may choose one.

SECONDARY OUTCOMES:
Most common referral process. Questionnaire | three months
  Participant may choose from the following options and choose more than one: Neurologist; GP; self-referral; MS nurse; other (please state); don't know
Most common provider of physiotherapy to the participant. Questionnaire | three months
  Participant may choose from the following options and choose more than one: NHS; private (self funded); private (insurance); charity; other (please state)
Most common physiotherapy intervention received for participant's MS. Questionnaire | three months
  Participant may choose form the following options and choose more than one: exercises to do at home prescribed by a physiotherapist; exercises with a physiotherapist; functional electrical stimulation, transcutaneous electrical stimulation; tilt table; acupuncture; advice or education from a physiotherapist; other (please state)
Most common pattern of physiotherapy appointments. Questionnaire | three months
  Participant may choose from the following options and choose only one: receiving physiotherapy sessions regularly; pattern varies depending on symptoms.
Most common expected waiting time from referral to receiving physiotherapy appointment. Questionnaire | three months
  Participant may choose form the following options and choose only one: less than a week; 1 to 2 weeks; 2 or more weeks but less than 4 weeks; 4 or more weeks but less than 6 weeks; 6 or more weeks but less than 12 weeks; 12 or more weeks.
Most common frequency of appointments. Questionnaire | three months
  Participant may choose form the following options and choose only one: once or more a week; once a fortnight; once every 1 to 3 months; twice a year; once a year or less
Most common length of physiotherapy sessions. Questionnaire | three months
  Participant may choose form the following options and choose only one: up to half an hour; between half an hour and an hour; more than an hour.
Most common number of people present at physiotherapy sessions. Questionnaire. | three months
  Participant may choose form the following options and choose more than one: one to one; 2- 4 people, 5 or more people; over the phone or internet.
Most common setting of receipt of physiotherapy. Questionnaire | three months
  Participant may choose form the following options and choose more than one: at home; in a hospital or clinic; in a community centre; in a charity centre; other (please state)
Number of participants who think they need more physiotherapy than they currently receive. Questionnaire | three months
  Participant may choose form the following options and choose only one: yes; no; don't know
Most common desired pattern of delivery of physiotherapy. Questionnaire | three months
  Participant may choose form the following options and choose only one: regularly; to vary depending on symptoms.
Most common desired frequency of appointments. Questionnaire | three months
  Participant may choose form the following options and choose only one: once or more a week; once a fortnight; once every 1 to 3 months; twice a year; once a year or less
Most common desired length of physiotherapy appointments. Questionnaire | three months
  Participant may choose form the following options and choose one: up to half an hour; between half an hour and an hour; more than an hour.
Most common desired setting for receiving physiotherapy. Questionnaire | three months
  Participant may choose form the following options and choose one: at home; in a hospital or clinic; in a community centre; in a charity centre; other (please state)
Most common desired number of people present at physiotherapy sessions. Questionnaire. | three months
  Participant may choose form the following options and choose one: one to one; 2- 4 people, 5 or more people; over the phone or internet.
Most common barriers to receiving physiotherapy. Questionnaire. | three months
  Participant may choose form the following options and choose more than one then rate their most severe from 1-3: Pain; fear of falling; bladder or bowels problems; fatigue; depression; anxiety/panic attacks; difficulty with walking; difficulty with wheelchair transfers; transport problems; distance to travel; lack of suitable parking; lack of time; family commitments; work commitments; cost; need someone to come with me; personal issues with physiotherapist; problems being referred to physiotherapy; physiotherapy is not available; physiotherapy will not be beneficial for me; there is nothing that makes it difficult for me to receive physiotherapy; other (please state)
Number of participants who have access to MS specialist services. Questionnaire | three months
  Participant may choose from the following options and choose one: yes; no.
Number of participants who are able to access MS specialist services as their needs change. Questionnaire | three months
  Participant may choose from the following options and choose one: yes; no.
Most common health professional available as part of MS specialist services. Questionnaire | three months
  Participant may choose from the following options and choose more than one: Occupational therapist; Social worker; MS specialist nurse; Continence nurse; Nurse: other (please state); Psychologist; GP; MS specialist Doctor/Neurologist; Doctor: other (please state); Speech and language therapist; Dietician; Orthotist; Other (please state)
Most commonly used health professional available as part of MS specialist services. Questionnaire | three months
  Participant may choose from the following options and choose more than one: Occupational therapist; Social worker; MS specialist nurse; Continence nurse; Nurse: other (please state); Psychologist; GP; MS specialist Doctor/Neurologist; Doctor: other (please state); Speech and language therapist; Dietician; Orthotist; Other (please state)
Number of participants who are offered a regular review for their MS. Questionnaire | three months
  Participant may choose from the following options and choose one: yes; no; don't know
Most common frequency of review. Questionnaire | three months
  Participant may choose from the following options and choose one: twice a year; once a year; less than once a year; don't know.
Most common health professional who carries out review. Questionnaire | three months
  Participant may choose from the following options and choose one: MS specialist Doctor/Neurologist; GP; Nurse; Physiotherapist; Occupational therapist; The person who does my review can vary; Other (please state)
Most common setting of review. Questionnaire | three months
  Participant may choose from the following options and choose one: at home; in a hospital or clinic; in a community centre; GP surgery; other (please state)
Most common disease modifying therapy taken in past. Questionnaire | three months
  Participant may choose from the following options and choose one: Beta-interferon (Rebif, Avonex, Betaferon); Glatiramer acetate (Copaxone); Dimethyl fumarate (Tecfidera); Teriflunomide (Aubagio); Natalizumab (Tysabri, Antigren); Fingolimod (Gilenya, Novartis); Mitoxantrone (novantrone); Alemtuzumab (Lemtrada); I have never taken any of these medications
Most common disease modifying therapy being taken. Questionnaire | three months
  Participant may choose from the following options and choose one: Beta-interferon (Rebif, Avonex, Betaferon); Glatiramer acetate (Copaxone); Dimethyl fumarate (Tecfidera); Teriflunomide (Aubagio); Natalizumab (Tysabri, Antigren); Fingolimod (Gilenya, Novartis); Mitoxantrone (novantrone); Alemtuzumab (Lemtrada); • I do not currently take any of these medications
Most commonly used complimentary therapy used for MS. Questionnaire | three months
  Participant may choose from the following options and choose more than one: Massage; Reflexology; Osteopathy or chiropractic; Magnet field therapy; The Alexander technique; Acupuncture or acupressure; Hyperbaric oxygen therapy; Reiki; Aromatherapy Relaxation or meditation; Homeopathy or herbal medicine; Other (please state)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Campbell, MRes, Principal Investigator — The University of Glasgow
Locations (1):
- The University of Glasgow, Glasgow, United Kingdom